CLINICAL TRIAL: NCT04398654
Title: Pulmonary Artery Sensor System Pressure Monitoring to Improve Heart Failure (HF) Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PASSPORT-HF
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Monitoring and therapy adjustment within the scope of the basic care described in the clinical trial plan.
- Intervention Group (Active Comparator): As in control group. In addition, in the intervention arm the CardioMEMSTM HF sensor implanted.
  Interventions: Device: CardioMEMSTM HF sensor - pulmonary artery pressure measurement

INTERVENTIONS:
Device: CardioMEMSTM HF sensor - pulmonary artery pressure measurement — CardioMEMSTM HF sensor implantation to meassure pulmonary artery pressure. Evaluation of the pressure curves by telemetric transmission and coordination of necessary adjustments of the therapy.
  Arms: Intervention Group

SUMMARY:
Randomized, parallel group controlled study examines the effect of supporting the Heart failure supply through pulmonary arterial (PA) pressure measurement with the CardioMEMS™ HF system to hard endpoints, safety and quality of life. The target population consists of heart failure (HF) patients who have been predominantly in New York Heart Association (NYHA) Stage III for the past 30 days and at least once in the past 12 months for HF were admitted to hospital. All patients receive basic care, which is based on structured telephone contact (between the care center, patient and family doctor) to optimize guideline compliant therapy. In the intervention group a PA pressure sensor is (CardioMEMS™-HF Sensor) implanted. These patients are structured by specially trained non-medical personnel aftercare with additional inclusion of the PA pressure values: adjusted to the basis of the information collected in PA monitoring the therapy is optimized. The follow-up period until the primary endpoint is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent received from the patient or a legal representative after the in-formation has been provided.
2. ≥≥ 18 years of age.
3. Predominant symptoms in NYHA Stage III in the 30-day period prior to consent to the study.
4. Objectified HF diagnosis for more than three months.
5. Hospitalisation within 12 months prior to inclusion due to deterioration of HF symptoms.
6. Able to tolerate dual antiplatelet therapy or anticoagulation therapy for one month after sensor implantation
7. Patients with reduced left ventricular ejection fraction (LVEF) ≤40% (diagnosed within 6 months prior to inclusion) must be treated with guideline-compliant HF pharmacotherapy; if one class of guideline-compliant medication is not tolerated, appropriate documentation must be supplied; patients must receive and tolerate at least one class of guideline-compliant medication; if no guideline-compliant medication is tolerated at all, the patient may not participate in the study.
8. In patients with preserved LVEF (>40%; diagnosed within 6 months prior to inclu-sion) comorbidities must be treated in accordance with guideline-compliant medi-cation.
9. Chest circumference (measured at axillary level) of less than 165 cm if BMI >35 kg/m2.
10. Willing and mentally and physically able to meet the requirements for follow-up and long-term basic care (this includes the long-term willingness of the patient, and of their relatives where relevant, to participate in PA pressure-based monitor-ing).
11. Appropriate domestic situation, defined as being accessible by telephone (via fixed or mobile network) .
12. For the intervention group: Implantation is only performed if the diameter of the pulmonary artery branch intended for implantation is ≥7 mm (assessment will be made during the right heart catheterization)

Exclusion criteria:

1. Enrolment in another study with an active treatment arm.
2. Severe cardiovascular event (e.g. myocardial infarction, open heart surgery, stroke, CRT implantation) in the 2 months prior to admission
3. Therapy-refractory heart failure in ACC/AHA stage D or new therapies that have taken place or are planned in the next 12 months (e.g. implantation of a left ven-tricular assist system / transplantation)
4. Active infection.
5. History of recurrent (>1 episode) pulmonary embolism and/or deep vein throm-bosis.
6. Continuous or intermittent chronic inotropic therapy.
7. Estimated glomerular filtration rate (eGFR) <25 ml/min
8. Life expectancy (according to the study physician's assessment) <12 months.
9. Severe, unrepaired congenital heart defect that would prevent implantation of the sensor.
10. Severe valve vitium with planned intervention in the next 3 months
11. Presence of a mechanical right heart valve.
12. Mental disorder that presumably (in the opinion of the study physician) has a negative impact on patient compliance or consent.
13. Failure of the coordinating physician to approve if the patient is enrolled in an HF disease management program or comparable case management program.
14. Women of childbearing age with a positive pregnancy test at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: composite of unplanned HF-related rehospitalisations and all-cause death | 12 months
  Composite endpoint of number of unplanned HF-related rehospitalisations or all-cause death
Primary safety endpoint: device-related complications | 12 months
  Rate of Device / System related complications
Co-primary safety endpoint: sensor failure | 12 months
  Rate of sensor failures

SECONDARY OUTCOMES:
Major secondary endpoint: changes in disease-related quality of life | 6 and 12 months
  Change in quality of life score after 6 and 12 month measured by Kansas City Cardiomyopathy questionnaire. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Changes in generic health-related quality of life | 6 and 12 months
  Change in Quality of Life score after 6 and 12 month measures by EQ-5D questionnaire.
  The EQ-5D-5L descriptive system comprises the five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), each dimension has five response levels:
  no problems, slight problems, moderate problems, severe problems, unable to /extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension (1 - 5, where higher scores indicate more severe problems).
  The EQ VAS records the respondent's overall current health on a vertical visual analogue scale (0-100), where the endpoints are labelled 'The best health you can imagine - 100' and 'The worst health you can imagine - 0'. The EQ VAS provides a quantitative measure of the patient's perception of their overall health.
HF-related mortality | 12 months
  Rate of HF-related mortality
Cardiovascular Mortality | 12 months
  Rate of cardiovascular mortality
All-cause Mortality | 12 months
  Rate of all-cause mortality
Unplanned HF-related hospitalizations | 12 months
  Rate of HF-related hospitalisations
Unplanned cardiovascular-related hospitalizations | 12 months
  Rate of cardiovascular-related hospitalisations
Unplanned all-cause hospitalizations | 12 months
  Rate of all-cause hospitalisations
Unplanned hospitalizations, other | 12 months
  Number of days alive and out of hospital
Non-serious Adverse Events | 12 months
  Rate of non-serious adverse events
Serious Adverse Events | 12 months
  Rate of serious adverse events
Symptoms of heart failure | 12 months
  Patient-reported symptoms of heart failure, measured by of the KCCQ Symptoms Score

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Störk, MD, Principal Investigator — Wuerzburg University Hospital
Locations (33):
- Germany (33):
  - SLK-Kliniken GmbH - Klinikum am Plattenwald, Bad Friedrichshall
  - Kerckhoff-Klinik Forschungs GmbH, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - BG Unfallkrankenhaus Berlin, Berlin
  - Charité Universitätsmedizin (Campus Mitte, Campus Benjamin Franklin), Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Praxis am Spreebogen, Berlin
  - Sana Klinikum Lichtenberg, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Coburg, Coburg
  - St. Vinzenz Hospital, Cologne
  - St Johannes Hospital Dortmund, Dortmund
  - Praxisklinik Herz und Gefäße, Dresden
  - St. Georg Klinikum, Eisenach
  - Helios Klinikum Erfurt, Erfurt
  - St. Elisabeth Krankenhaus, Contilia Herz- und Gefäßzentrum, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Gießen, Giessen
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Westpfalz Klinikum, Kaiserslautern
  - Klinikum Karlsburg, Karlsburg
  - Leipzig Heart Institute GmbH, Leipzig
  - Cardio Centrum Ludwigsburg-Bietigheim, Ludwigsburg
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Vest, Recklinghausen
  - Cardio Consil Rostock, Rostock
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Rems-Murr Klinikum, Winnenden
  - Deutsches Zentrum für Herzinsuffizienz (DZHI), Würzburg

REFERENCES:
- [Derived] Stork S, Bernhardt A, Bohm M, Brachmann J, Dagres N, Frantz S, Hindricks G, Kohler F, Zeymer U, Rosenkranz S, Angermann C, Assmus B. Pulmonary artery sensor system pressure monitoring to improve heart failure outcomes (PASSPORT-HF): rationale and design of the PASSPORT-HF multicenter randomized clinical trial. Clin Res Cardiol. 2022 Nov;111(11):1245-1255. doi: 10.1007/s00392-022-01987-3. Epub 2022 Mar 4. PMID 35246723